CLINICAL TRIAL: NCT04154852
Title: Prospective, Single-centre, Double-Blind, Randomised, Placebo-controlled Study Evaluating Efficacy of Adalimumab + Methotrextate Compared With Placebo + Methotrexate in Patients With Early Oligoarthritis (ADEOS)
Brief Title: ADalimumab in Persistent Early Oligoarthrits Study (ADEOS)
Acronym: ADEOS
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Leeds (Other)
Collaborators: Abbott (Industry)
Responsible Party: Principal Investigator, Dr Ai Lyn Tan, Chief Investigator, University of Leeds
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: RR08/8685; 2008-004877-17 (EudraCT Number); 10060 (Other: UKCRN)
Record Dates: First submitted 2014-04-15; First posted 2019-11-07 (Actual); Last update posted 2019-11-07 (Actual); Status verified 2019-11

CONDITIONS: Oligoarthritis
MeSH Terms: conditions — Arthritis | interventions — Adalimumab; Methotrexate; Folic Acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- TNF-antagonist (Experimental): Adalimumab, 40 mg, 2-weekly Methotrexate, rapid escalation to 25mg, weekly Folic Acid 5mg, 6 days a week
  Interventions: Drug: Adalimumab; Drug: Methotrexate; Drug: Folic Acid
- Placebo + MTX (Active Comparator): Placebo, 2 weekly Methotrexate, rapid escalation to 25mg, weekly Folic Acid 5mg, 6 days a week
  Interventions: Drug: Methotrexate; Drug: Placebo; Drug: Folic Acid

INTERVENTIONS:
Drug: Adalimumab
  Arms: TNF-antagonist
Drug: Methotrexate
Drug: Placebo — Placebo to replace adalimumab
  Arms: Placebo + MTX
Drug: Folic Acid

SUMMARY:
The purpose of this study is to investigate adalimumab, a drug that is currently licensed for treatment of patients with rheumatoid arthritis, psoriatic arthritis, ankylosing spondylitis and inflammatory bowel disease (Crohn's disease). It is a protein (human monoclonal antibody) that is designed to block the effects of an inflammatory cytokine, tumour necrosis factor alpha (TNF alpha) which is a causative factor in joint inflammation. It is given as a subcutaneous injection.

Management of established rheumatoid arthritis has been transformed with the use of TNFantagonists, the first in the class of biological agents. The benefits in early RA are also continuing to emerge. Oligoarthritis represents a subgroup of early inflammatory arthritis that warrants more effective treatment strategy including the potential to modulate the disease course and halt further progression. The TNFantagonists offer the potential of achieving this, justifying this initial investigation.

Hence, this study is designed to establish the benefit of adalimumab in preventing progression of oligoarthritis. The primary aim of the study is to assess how many patients achieve remission i.e. no further evidence of joint inflammation or damage. The investigators will do this by including patients who present with inflammation of four or less joints who do not fulfil criteria for a definite arthritis condition such as rheumatoid arthritis. The investigators will perform clinical, laboratory (blood tests) and imaging assessments at regular intervals on these patients to check on safety of the study drug adalimumab and evaluate any changes in disease activity that may have resulted from use of adalimumab. All patients will receive treatment with a standard therapy (methotrexate) with randomisation of half of the patients to receive the active study drug, adalimumab as additional treatment for six months.

ELIGIBILITY:
Inclusion Criteria:

Subjects presenting at the rheumatology clinic who meet all of the following criteria will be considered for enrolment into the study:-

* Male and female patients aged between 18 and 80 years.
* Oligoarthritis defined as inflammatory arthritis affecting ≤ 4 joints
* At least 1 large joint involvement (wrist, elbow, shoulder, knee or ankle)
* Disease duration of less than 12 months
* Patients on NSAIDs must have remained on an unchanged regimen for at least 28 days prior to study drug administration.
* Patients must be able and willing to comply with the terms of this protocol.
* Informed consent must be obtained in writing for all subjects at enrolment into the study.

Exclusion Criteria:

* Patients who have > 12 months disease duration
* Exclude if DIP joint alone
* Evidence of osteoarthritis
* Diagnosis of gout
* Previous treatment with a DMARD therapy.
* Change in NSAID dose within the last 28 days
* Previous treatment with oral, intra-muscular or intra-articular steroid
* Patients unwilling or unable to receive adalimumab or MTX or both for the duration of the study.
* Planned surgery within 12 months of study initiation.
* Patients with moderate to severe heart failure
* Suspicion of diagnosis of tuberculosis (positive tuberculosis test (>5mm in duration if previous BCG or >10mm if no previous BCG) or abnormal chest x-ray)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2011-06; Primary Completion 2017-01-16 (Actual); Study Completion 2017-01-16 (Actual)

PRIMARY OUTCOMES:
Patients in remission at 24 weeks. | 24 weeks
  Number in remission at 24 weeks (absence of clinical-evidence synovitis (no tender/swollen joints) & CRP< 5mg/ml)

SECONDARY OUTCOMES:
Complete response at weeks 12, 36, 48, 72 and 96 | Weeks 12, 36, 48, 72 and 96.
  Complete response (absence of clinical-evidence synovitis & CRP< 5mg/ml) at weeks 12, 36, 48, 72 and 96
Disease Activity Score at weeks 12, 24, 36, 48, 72 and 96 | Weeks 12, 24, 36, 48, 72 and 96
  Disease Activity Score at weeks 12, 24, 36, 48, 72 and 96
Ultrasonographical features (erosions) at weeks 2 and 24 | Week 2 and 24
  Ultrasonographical features (erosions) at weeks 2 and 24
Health Assessment Questionnaire at weeks 0, 12 24, 36, 48, 72 and 96 | Week 0, 12 24, 36, 48, 72 and 96
  Health Assessment Questionnaire at weeks 0, 12 24, 36, 48, 72 and 96
EQ-5D (Euro-QoL) questionnaire at weeks 0, 12 24, 36, 48, 72 and 96 | Week 0, 12 24, 36, 48, 72 and 96
  EQ-5D (Euro-QoL) questionnaire at weeks 0, 12 24, 36, 48, 72 and 96
Work Instability Scale at weeks 0, 12, 24, 36, 48, 72 and 96 | weeks 0, 12, 24, 36, 48, 72 and 96
  Work Instability Scale at weeks 0, 12, 24, 36, 48, 72 and 96
Plain radiography at weeks -2, 24 and 96 | weeks -2, 24 and 96
  Plain radiography at weeks -2, 24 and 96

CONTACTS AND LOCATIONS:
Overall Officials: Dr Ai Lyn Tan, Principal Investigator — University of Leeds
Locations (1):
- Leeds Teaching Hospitals NHS Trust, Leeds, West Yorkshire, United Kingdom